CLINICAL TRIAL: NCT01733563
Title: Effects of Carbohydrate Containing Diets on Lipid Metabolism & Fatty Acid Oxidation in Healthy Young Men - a Randomized, Double-Blinded Study.
Brief Title: Sugar Sweetened Beverages (SSB)- Effects on Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: SNF Swiss National Foundation (Unknown); University of Lausanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SSB-Effects on metabolism
Record Dates: First submitted 2012-11-09; First posted 2012-11-27 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Metabolism
Keywords: sugar sweetened beverages; fructose; lipogenesis; beta-oxidation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- fructose sweetened beverage (Experimental): Soft drink consumption:
  Subjects have to drink a fructose sweetened beverage (3x 200ml per day, 13.3g fructose/100ml) during 7 weeks
  Interventions: Procedure: Soft drink consumption
- glucose sweetened beverage (Experimental): Soft drink consumption:
  Subjects have to drink a glucose sweetened beverage (3x 200ml per day, 13.3g glucose/100ml) during 7 weeks
  Interventions: Procedure: Soft drink consumption
- sucrose sweetened beverage (Experimental): Soft drink consumption:
  Subjects have to drink a sucrose sweetened beverage (3x 200ml per day, 13.3g sucrose/100ml) during 7 weeks
  Interventions: Procedure: Soft drink consumption
- No change of eating habits (Experimental): No Soft drink consumption (no soft drink diet):
  Subjects do not change their eating habits during 7 weeks
  Interventions: Procedure: Soft drink consumption

INTERVENTIONS:
Procedure: Soft drink consumption

SUMMARY:
The objective of this study is to investigate the impact of sugar sweetened beverages on the fat metabolism of healthy young men. It is well known that consumption of beverages sweetened with fructose is associated with different health risks such as type 2 diabetes. The present study has been designed to dissect differences in the metabolic pathways of fructose and glucose, but also metabolic adaptations during fructose, glucose and sucrose diets. During a period of seven weeks subjects will consume either fructose, glucose or sucrose sweetened beverages or continue their usual drinking habits. During these seven weeks there will be different metabolic investigations using stable isotope tracers. First, the rate of lipolysis and beta-oxidation will be determined. Second, the rates of fatty acid synthesis will be measured. During all examinations there will also be substrate- and energy-utilization measurements by indirect calorimetry, blood analysis and morphometric measurements. Based on the literature main hypotheses are: Fructose enhances de novo lipogenesis postprandially and also in the fasting state significantly more than glucose by enhanced expression of lipogenic enzymes. Fructose decreases beta oxidation via downregulation of oxidative enzymes.

ELIGIBILITY:
Inclusion criteria:

* Healthy male volunteers aged 18-30
* BMI between 19-24 kg/m2
* Non-smoker

Exclusion criteria:

* Acute or chronic infections, malignant disease, renal, hepatic (more than two-fold increased transaminases), pulmonary, neurological (epilepsy) or psychiatric diseases, manifested atherosclerosis, or any other disease precluding participation in the study.
* Diabetes
* Known alcohol, substance or drug abuse, concomitant medication
* More than three hours of physical exercise per week
* Consumption of more than 2 times 3 dl SSB daily
* Subjects likely to fail to comply with the study protocol
* Subjects who do not give informed consent

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Lipogenesis | After total 6 weeks dietary intervention
  Measurement of lipogenesis is based on i. v. administration of stable isotope labelled acetate (1,2-13C-acetate). 13C incorporation into palmitate is quantified by mass-spectrometry. 13C incorporation correlates to the rate of fatty acid synthesis.

SECONDARY OUTCOMES:
Lipolysis | After total 6 weeks dietary intervention
  Measurements using stable isotopes

OTHER OUTCOMES:
Waist/Hip Ratio | After total 6 weeks dietary intervention
  Measurement waist/hip ratio using a nonstretchable band

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Gerber, MD, Principal Investigator — University Hospital Zurich, Endocrinology and Diabetology
Locations (1):
- University Hospital Zurich, Endocrinology and Diabetology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Geidl-Flueck B, Hochuli M, Nemeth A, Eberl A, Derron N, Kofeler HC, Tappy L, Berneis K, Spinas GA, Gerber PA. Fructose- and sucrose- but not glucose-sweetened beverages promote hepatic de novo lipogenesis: A randomized controlled trial. J Hepatol. 2021 Jul;75(1):46-54. doi: 10.1016/j.jhep.2021.02.027. Epub 2021 Mar 6. PMID 33684506